CLINICAL TRIAL: NCT03102177
Title: Hypothyroidism Treatment in Aging and Thyroid Cancer
Brief Title: Effect of Age, Weight and Sex on Levothyroxine Pharmacokinetics
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010-572
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hypothyroidism Primary
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: Open label prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stable isotope arm (Experimental): Measurement of blood levels of labelled levothyroxine after administration of single oral dose of stable isotope levothyroxine
  Interventions: Drug: Administration of stable Isotope labeled levothyroxine

INTERVENTIONS:
Drug: Administration of stable Isotope labeled levothyroxine — Administration of single dose of stable isotope carbon-13 labeled levothyroxine and measurement of blood levels of stable isotope-labeled levothyroxine
  Other Names: levothyroxine or synthroid

SUMMARY:
This study was a prospective, single-center, open-label, non-randomized, pharmacokinetic study using stable isotope carbon-13 labeled levothyroxine

DETAILED DESCRIPTION:
Setting The study was conducted on the clinical research unit of an academic medical center.

Participants Adults of any age being treated with levothyroxine for hypothyroidism were studied.

Interventions A single dose of 13C- LT4 was administered to hypothyroid subjects taking levothyroxine replacement.

Main Outcomes and Measures Eighteen serial plasma samples were collected. One sample was obtained before the 13C- LT4 dose and the remainder over the 312-hour period post-dosing. 13C- LT4 concentration was quantified using validated liquid chromatography tandem mass spectrometry methods. Pharmacokinetic analysis was conducted using linear log trapezoidal non-compartmental analysis using Phoenix 6.4.

ELIGIBILITY:
Inclusion Criteria:

* age >21 years at the time of consent
* euthyroidism while undergoing treatment with LT4
* no other serious illness
* ability to give written informed consent.

Exclusion Criteria:

* baseline hematocrit lower than 28.0%
* TSH greater than 4.5 mIU/L
* kidney dysfunction
* concomitant use of drugs that affect thyroidal axis interactions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
CL/F | 120 hours
  oral clearance rate (defined as the ratio of dose administered to AUC0-∞)
V/F | 120 hours
  apparent volume of distribution (estimated by CL/F/ λ)
t-half | 120 hours
  the half-life of the terminal disposition phase (t-half) estimated by ln(2)/λ .

SECONDARY OUTCOMES:
CL/F analysed by age groups | 120 hours
  CL/F will be compared in adults (age ≤60 years) versus elderly (age>60 years) using Wilcoxon signed-rank test using significance level of α = 0.05. Additionally, these PK parameters were regressed against age (as a continuous covariate).
  Sex (male or female), weight (as a continuous covariate), and body mass index (BMI) (as a continuous covariate) will be considered using a stepwise linear regression approach.
V/F analysed by age groups | 120 hours
  V/F will be compared in adults (age ≤60 years) versus elderly (age>60 years) using Wilcoxon signed-rank test using significance level of α = 0.05. Additionally, these PK parameters were regressed against age (as a continuous covariate).
  Sex (male or female), weight (as a continuous covariate), and body mass index (BMI) (as a continuous covariate) will be considered using a stepwise linear regression approach.
t-half by age groups | 120 hours
  t-half will be compared in adults (age ≤60 years) versus elderly (age>60 years) using Wilcoxon signed-rank test using significance level of α = 0.05. Additionally, these PK parameters were regressed against age (as a continuous covariate).
  Sex (male or female), weight (as a continuous covariate), and body mass index (BMI) (as a continuous covariate) will be considered using a stepwise linear regression approach.

IPD SHARING:
Plan to Share IPD: No